CLINICAL TRIAL: NCT03055013
Title: A Phase 3 RandOmized Study Comparing PERioperative Nivolumab vs. Observation in Patients With Renal Cell Carcinoma Undergoing Nephrectomy (PROSPER RCC)
Brief Title: Nivolumab in Treating Patients With Localized Kidney Cancer Undergoing Nephrectomy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCI-2016-00326; NCI-2016-00326 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA8143; EA8143 (Other: ECOG-ACRIN Cancer Research Group); EA8143 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2017-02-15; First posted 2017-02-16 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Renal Cell Carcinoma; Sarcomatoid Renal Cell Carcinoma; Stage II Renal Cell Cancer AJCC v7; Stage III Renal Cell Cancer AJCC v7; Unclassified Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nephrectomy; Nivolumab; Watchful Waiting; Observation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (nivolumab + nephrectomy) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 14 days for 2 cycles. Patients then undergo partial or radical nephrectomy 7-28 days later. Patients then receive nivolumab over 30 IV on day 1. Treatment repeats every 14 days for 6 cycles, and then every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Patients enrolled after Amendment 4 receive nivolumab IV over 30 minutes on day 1. Patients then undergo partial or radical nephrectomy 7-28 days later. Patient then receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 4 weeks for up to 9 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Nephrectomy; Biological: Nivolumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (nephrectomy only) (Active Comparator): Patients undergo partial or radical nephrectomy within 8 weeks after registration followed by observation.
  Interventions: Procedure: Nephrectomy; Other: Patient Observation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Nephrectomy — Undergo nephrectomy
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm A (nivolumab + nephrectomy)
Other: Patient Observation — Undergo observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Arm B (nephrectomy only)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares nephrectomy (surgery to remove a kidney or part of a kidney) with nivolumab to the usual approach of nephrectomy followed by standard post-operative follow-up and monitoring, in treating patients with kidney cancer that is limited to a certain part of the body (localized). Nivolumab is a drug that may help stimulate the immune system to attack any cancer cells that may remain after surgery. The addition of nivolumab to the usual surgery could prevent the cancer from returning. It is not yet known whether nivolumab and nephrectomy is more effective than nephrectomy alone in treating patients with kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare recurrence-free survival (RFS) between patients with renal cell carcinoma randomly assigned to perioperative nivolumab in conjunction with radical or partial nephrectomy with patients randomized to surgery alone.

SECONDARY OBJECTIVES:

I. To evaluate for differences in recurrence-free survival associated with perioperative nivolumab compared to surgery alone among the subset of patients with clear cell histology.

II. To compare the overall survival between the two arms. III. To describe the safety and tolerability of perioperative nivolumab.

CORRELATIVE OBJECTIVES:

I. To correlate the primary tumor's expression of PD-L1 with outcome. II. To correlate the expression of PD-L1 on tumor tissue at nephrectomy and recurrence with outcome.

III. To archive images for potential central confirmation of recurrence and for future correlative work with American College of Radiology Imaging Network (ACRIN), including markers predicting outcome or response.

IV. To prospectively collect tumor and biologic specimens (e.g., serum, peripheral blood mononuclear cells [PBMCs]) for future correlative studies.

V. To characterize the pharmacokinetics of nivolumab and explore exposure response relationships with respect to safety and efficacy.

VI. To characterize the immunogenicity of nivolumab.

QUALITY OF LIFE OBJECTIVE:

I. To evaluate differences in change from baseline in patient-reported symptoms and toxicities among patients randomized to treatment with nivolumab compared to surgery alone.

OTHER EXPLORATORY OBJECTIVES:

I. To explore descriptively the efficacy of treatment with nivolumab in patients with non-clear cell (including unclassified) histologies.

II. To characterize the effects of nivolumab on bone metabolism and bone density.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 14 days for 2 cycles. Patients then undergo partial or radical nephrectomy 7-28 days later. Patient then receive nivolumab over 30 IV on day 1. Treatment repeats every 14 days for 6 cycles, and then every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

Patients enrolled after Amendment 4 receive nivolumab IV over 30 minutes on day 1. Patients then undergo partial or radical nephrectomy 7-28 days later. Patients then receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 4 weeks for up to 9 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients undergo partial or radical nephrectomy within 8 weeks after registration followed by observation.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and every 12 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY CRITERIA FOR RANDOMIZATION:
* Patients must have a renal mass consistent with a clinical stage >= T2Nx renal cell carcinoma (RCC) or TanyN+ RCC for which radical or partial nephrectomy is planned
* Patients must have no clinical or radiological evidence of distant metastases (M0) unless the presumed M1 disease is planned to be resected/definitively treated (e.g., thermal ablation, stereotactic radiation) at the same time or up to 12 weeks after the date of the initial procedure such that the patient is considered "no evidence of disease" (M1 NED)

  * Liver, bone, or brain metastases are not permitted
  * No more than 3 metastases are permitted, and all must be able to be removed or definitively treated within 12 weeks of the primary tumor resection
* If histological confirmation of RCC has not been done within 12 months prior to randomization, patient must be willing to undergo a core biopsy for this purpose if randomized to Arm A

  * NOTE: This histologic confirmation can be a (1) standard of care diagnostic biopsy or (2) a research biopsy or a planned metastasectomy. Tissue must be obtained with results available prior to the neoadjuvant dose

    * Patients randomized to Arm A: core tumor biopsy must have demonstrated RCC of any histology, including sarcomatoid, unclassified, or "unknown histology" (if preoperative biopsy was uninformative) with exception below for non-diagnostic biopsies
    * If the biopsy performed following randomization clearly demonstrates a benign condition, oncocytoma or a different type of cancer that is not RCC, the patient is not eligible and must come off study
    * A non-diagnostic biopsy is considered a good faith effort and does not need to be repeated unless deemed clinically necessary by the treating investigator
* Patient must not have any prior systemic or local anti-cancer therapy for the current RCC

  * Patient must not have undergone a partial nephrectomy for the current RCC
  * Patient must not have had a metastasectomy for the current RCC diagnosis unless performed to render patient NED (in addition to the planned nephrectomy) within 6 months prior to the current diagnosis
  * Patient must not have received current or past antineoplastic systemic therapies for RCC: i.e., chemotherapy, hormonal therapy, immunotherapy, or standard or investigational agents for treatment of RCC
  * Patient must not have received prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Patient must be >= 18 years of age. Because no dosing or adverse event data are currently available on the use of nivolumab therapy in patients < 18 years of age, children are excluded from this study
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patient must not have a prior history of RCC that was treated with curative intent within the past 5 years

  * Patients with a prior RCC that was treated > 5 years before, are eligible if the current tumor is consistent with a new primary in the opinion of the treating investigator
  * Patients with bilateral synchronous RCCs are eligible if they can be resected or definitively treated at the same time or within a 12 week window from time of initial nephrectomy (partial or radical) or procedure and maintain adequate residual renal function; the patient is not eligible if both kidneys are to be completely removed and subsequent hemodialysis will be required

    * Permitted forms of local therapy for second tumor:

      * Partial or radical nephrectomy
      * If kidney tumor is =< 3 cm: thermal ablation (e.g., radiofrequency ablation, cryoablation or stereotactic radiosurgery)
* Patients cannot have concurrent malignancies, with the following exceptions:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer

    * A history of superficial Ta urothelial cancer is permitted (as long as not currently undergoing treatment) whereas T1 or greater disease is excluded if < 3 years from diagnosis; concurrent persistent disease is not permitted
    * Adequately treated stage I or II cancer from which the patient is currently in complete remission
    * Any other cancer and stage from which the patient has been disease-free for at least 3 years prior to the time of randomization and as long as they are not receiving any current treatment (e.g. adjuvant or maintenance systemic or local therapy)
    * Concurrent low risk prostate cancer on active surveillance
* Patient must not have active known or suspected autoimmune disease. The following autoimmune disorders are permitted: patients with vitiligo, type I diabetes mellitus, controlled/stable hypo or hyperthyroidism due to autoimmune or non-autoimmune conditions (hormone replacement is allowed), psoriasis not requiring systemic treatment, or other conditions not expected to recur
* Patient must not have any ongoing condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications with the exceptions outlined below; patient must not have received any treatment with other immunosuppressive agents within 14 days prior to the first dose of study drug with the following exceptions:

  * Topical, ocular, intra-articular, intranasal, inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone or the equivalent are permitted in the absence of active autoimmune disease
  * A brief (less than 3 weeks) course of corticosteroids (any amount) for prophylaxis (for example: contrast dye allergy) or for treatment of non-autoimmune conditions (for example: nausea, delayed-type hypersensitivity reaction caused by a contact allergen) is permitted
* Patient must not have uncontrolled adrenal insufficiency
* Patient must not have known evidence of chronic active liver disease or evidence of acute or chronic hepatitis B Virus (HBV) or hepatitis C (HCV); HBV and HCV testing must be completed within 8 weeks prior to randomization

  * NOTE: If the patient has been treated and cured, and the HCV ribonucleic acid (RNA) is undetectable, the patient is eligible for this study
* Patient must not have any serious intercurrent illness, including ongoing or active infection requiring parenteral antibiotics
* Patient must not have known evidence of human immunodeficiency virus (HIV) infection, since the effects of nivolumab on anti-retroviral therapy have not been studied; HIV testing is only required if past or current history is suspected
* Patient must not have any known medical condition (e.g. a condition associated with uncontrolled diarrhea such as ulcerative colitis or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or interfere with the interpretation of safety results
* Patient must not have had any major surgery within 28 days prior to randomization
* Patient must not be currently enrolled in other clinical trials testing a therapeutic intervention
* Patient must not have any history of severe hypersensitivity to a monoclonal antibody
* Patient must have the ability to understand and the willingness to sign a written informed consent document
* Patients must not be pregnant or breast-feeding, as the effects of nivolumab on the developing human fetus or in the nursing infant are unknown; all patients of childbearing potential must have a blood test or urine study within 2 weeks prior to randomization to rule out pregnancy; a patient of childbearing potential is defined as any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patients must not expect to conceive or father children by using accepted and effective method(s) of contraception, as described in the informed consent form (ICF), or by abstaining from sexual intercourse for the duration of their participation in the study; patients of childbearing potential must use adequate methods to avoid pregnancy for 5 months after the last dose of nivolumab
* White blood cells >= 2000/uL (within 8 weeks prior to randomization)
* Absolute neutrophil count (ANC) >= 1,500/mm^3 (within 8 weeks prior to randomization)
* Platelet count >= 100,000/mm^3 (within 8 weeks prior to randomization)
* Hemoglobin >= 9.0 g/dL (within 8 weeks prior to randomization)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or calculated creatinine clearance (CrCl) >= 40mL/min (within 8 weeks prior to randomization)
* Total bilirubin =< 1.5 x ULN (except subjects with Gilbert syndrome, who can have total bilirubin < 3.0 x ULN) (within 8 weeks prior to randomization)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN (within 8 weeks prior to randomization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 819 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2031-06-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Harshman, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (414):
- United States (397):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Veterans Administration Medical Center - Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Community Cancer Institute, Clovis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - The Watson Clinic, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Albany Medical Center, Albany, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Rex Hematology Oncology Associates-Cary, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Rex Hematology Oncology Associates-Blue Ridge, Raleigh, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - UNC Rex Cancer Center of Wakefield, Raleigh, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (15):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Saint Joseph's Healthcare Charlton Campus, Hamilton, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Niagara Health System-Saint Catharines General, Saint Catharines, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
- Israel (2):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem

REFERENCES:
- [Derived] Allaf ME, Kim SE, Master V, McDermott DF, Harshman LC, Cole SM, Drake CG, Signoretti S, Akgul M, Baniak N, Li-Ning E, Palmer MB, Emamekhoo H, Adra N, Kaimakliotis H, Ged Y, Pierorazio PM, Abel EJ, Bilen MA, Ogan K, Moon HH, Ramaswamy KA, Singer EA, Mayer TM, Lohrey J, Margulis V, Gills J, Delacroix SE, Waples MJ, James AC, Wang P, Choueiri T, Michaelson MD, Kapoor A, Heng DY, Shuch B, Leibovich BC, Lara PN, Manola J, Maskens D, Battle D, Uzzo R, Bratslavsky G, Haas NB, Carducci MA. Perioperative nivolumab versus observation in patients with renal cell carcinoma undergoing nephrectomy (PROSPER ECOG-ACRIN EA8143): an open-label, randomised, phase 3 study. Lancet Oncol. 2024 Aug;25(8):1038-1052. doi: 10.1016/S1470-2045(24)00211-0. Epub 2024 Jun 25. PMID 38942046
- [Derived] Marconi L, Sun M, Beisland C, Klatte T, Ljungberg B, Stewart GD, Dabestani S, Choueiri TK, Bex A. Prevalence, Disease-free, and Overall Survival of Contemporary Patients With Renal Cell Carcinoma Eligible for Adjuvant Checkpoint Inhibitor Trials. Clin Genitourin Cancer. 2021 Apr;19(2):e92-e99. doi: 10.1016/j.clgc.2020.12.005. Epub 2021 Jan 7. PMID 33526329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on February 2, 2017 and closed to accrual on June 2, 2021, with a total enrollment of 819 patients.
Groups:
- Arm A (Nephrectomy + Nivolumab): Patients receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 14 days for 2 cycles. Patients then undergo partial or radical nephrectomy 7-28 days later. Patients then receive nivolumab over 30 IV on day 1. Treatment repeats every 14 days for 6 cycles, and then every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Patients enrolled after Amendment 4 receive nivolumab IV over 30 minutes on day 1. Patients then undergo partial or radical nephrectomy 7-28 days later. Patient then receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 4 weeks for up to 9 cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Nephrectomy + Nivolumab) | Arm B (Nephrectomy Only)
Started | 404 | 415
RCC Patients | 381 | 399
Patients Who Received Treatment and Were Assessed for Adverse Events | 357 | 377
Completed | 197 | 387
Not Completed | 207 | 28
Not completed — Adverse Event | 78 | 0
Not completed — Death | 6 | 0
Not completed — Disease relapse | 33 | 0
Not completed — Withdrawal by Subject | 28 | 0
Not completed — Other complicating disease | 5 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Benign mass/non-RCC | 4 | 0
Not completed — Enrolled in another trial | 1 | 0
Not completed — Non-protocol therapy | 1 | 0
Not completed — Incompliance | 1 | 0
Not completed — Insurance issues | 1 | 0
Not completed — Did not receive nivolumab and surgery | 38 | 0
Not completed — Did not receive nivolumab | 10 | 0
Not completed — Did not receive surgery | 0 | 28

BASELINE CHARACTERISTICS:
Population: All randomized RCC patients are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Nephrectomy + Nivolumab) | Arm B (Nephrectomy Only) | Total
Number analyzed (Participants) | 381 | 399 | 780
Age, Continuous [Median (Full Range); unit: years] | 60 [31 to 88] | 61 [23 to 88] | 61 [23 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 122 | 235
  Male | 268 | 277 | 545
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 34 | 73
  Not Hispanic or Latino | 333 | 352 | 685
  Unknown or Not Reported | 9 | 13 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 13 | 11 | 24
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 30 | 29 | 59
  White | 311 | 326 | 637
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 24 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival (RFS) Rate at 5 Years
Description: RFS is defined as time from randomization to disease recurrence or death from any cause. Patients who did not undergo nephrectomy or were not disease-free following nephrectomy were considered as having an event at day 1. Patients that are alive without an event were censored at the date of last disease evaluation. RFS rate at 5 years was the proportion of patients who are recurrence-free and alive at 5 years based on Kaplan-Meier estimates.
Time Frame: Assessed at 20 weeks, 40 weeks, then every 3 months for patients <2 years from randomization, then every 6 months for 3 years
Population: All randomized RCC patients were included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Nephrectomy + Nivolumab) | Arm B (Nephrectomy Only)
Number analyzed (Participants) | 381 | 399
proportion of participants | 0.63 [0.577 to 0.688] | 0.605 [0.545 to 0.671]
Statistical Analysis 1: Comparison: Arm A (Nephrectomy + Nivolumab) vs Arm B (Nephrectomy Only); Test type: Superiority; p = 0.34, Log Rank; stratified logrank test (one-sided); Cox Proportional Hazard = 0.95, 95% CI 2-sided [0.74 to 1.22] — hazard ratio : arm A vs. arm B

2. Secondary Outcome: Recurrence-free Survival (RFS) Rate at 3 Years Among Patients With Clear Cell Histology
Description: RFS is defined as time from randomization to disease recurrence or death from any cause. Patients who did not undergo nephrectomy or were not disease-free following nephrectomy were considered as having an event at day 1. Patients that are alive without an event were censored at the date of last disease evaluation. RFS rate at 3 years was the proportion of patients who are recurrence-free and alive at 3 years based on Kaplan-Meier estimates.
Time Frame: Assessed at 20 weeks, 40 weeks, then every 3 months for patients <2 years from randomization, then every 6 months for 1 year
Population: All randomized RCC patients who had clear cell histology according to surgery or biopsy were included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Nephrectomy + Nivolumab) | Arm B (Nephrectomy Only)
Number analyzed (Participants) | 303 | 325
proportion of participants | 0.663 [0.606 to 0.725] | 0.675 [0.623 to 0.732]

3. Secondary Outcome: Overall Survival Rate at 5 Years
Description: Overall survival is defined as time from randomization to death from any cause. Overall survival rate at 5 years was the proportion of patients who are alive at 5 years based on Kaplan-Meier estimates.
Time Frame: as for outcome 1
Population: All randomized patients were included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Nephrectomy + Nivolumab) | Arm B (Nephrectomy Only)
Number analyzed (Participants) | 404 | 415
proportion of participants | 0.73 [0.611 to 0.873] | 0.811 [0.728 to 0.904]

4. Other Pre Specified Outcome: Association Between the Primary Tumor's Expression of PD-L1 With Outcome
Description: Association between the primary tumor's expression of PD-L1 with outcome
Time Frame: Assessed at 20 weeks, 40 weeks, then every 3 months for patients <2 years from randomization, then every 6 months for 3 years, then annually for 5 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Association Between the Expression of PD-L1 on Tumor Tissue at Nephrectomy as Well as Recurrence and Outcome
Description: Association between the expression of PD-L1 on tumor tissue at nephrectomy as well as recurrence and outcome
Time Frame: as for outcome 4
Reporting Status: Not Posted

6. Other Pre Specified Outcome: To Archive Images for Potential Central Confirmation of Recurrence and for Future Correlative Work
Description: To archive images for potential central confirmation of recurrence and for future correlative work
Time Frame: as for outcome 4
Reporting Status: Not Posted

7. Other Pre Specified Outcome: To Collect Tumor and Biologic Specimens for Future Correlative Studies
Description: To collect tumor and biologic specimens for future correlative studies
Time Frame: Assessed at baseline, nephrectomy, 9 months and recurrence
Reporting Status: Not Posted

8. Other Pre Specified Outcome: To Characterize the Pharmacokinetics of Nivolumab and Explore Exposure Response Relationships With Respect to Safety and Efficacy
Description: To characterize the pharmacokinetics of nivolumab and explore exposure response relationships with respect to safety and efficacy
Time Frame: as for outcome 4
Reporting Status: Not Posted

9. Other Pre Specified Outcome: To Characterize the Immunogenicity of Nivolumab
Description: To characterize the immunogenicity of nivolumab
Time Frame: as for outcome 4
Reporting Status: Not Posted

10. Other Pre Specified Outcome: To Evaluate Differences in Change From Baseline in Patient-reported Symptoms and Toxicities Among Patients Randomized to Treatment With Nivolumab Compared to Surgery Alone
Description: To evaluate differences in change from baseline in patient-reported symptoms and toxicities among patients randomized to treatment with nivolumab compared to surgery alone
Time Frame: Assessed at baseline, pre-nephrectomy, 8 weeks post-nephrectomy, 20 weeks, 40 weeks, 54 weeks, recurrence and 2 years post randomization
Reporting Status: Not Posted

11. Other Pre Specified Outcome: To Explore Descriptively the Efficacy of Treatment With Nivolumab in Patients With Non-clear Cell (Including Unclassified) Histologies.
Description: To explore descriptively the efficacy of treatment with nivolumab in patients with non-clear cell (including unclassified) histologies.
Time Frame: as for outcome 4
Reporting Status: Not Posted

12. Other Pre Specified Outcome: To Characterize the Effects of Nivolumab on Bone Metabolism and Bone Density
Description: To characterize the effects of nivolumab on bone metabolism and bone density
Time Frame: as for outcome 4
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, up to 6 years
Description: All patients registered on this study were included in the all-cause mortality analysis. Patients who received treatment and were assessed for adverse events were included in the analysis of adverse events.
Arm/Group | Arm A (Nephrectomy + Nivolumab) | Arm B (Nephrectomy Only)
All-Cause Mortality (participants affected / at risk) | 48/404 | 40/415
Serious Adverse Events (participants affected / at risk) | 113/357 | 46/377
Other Adverse Events (participants affected / at risk) | 278/357 | 114/377
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Nephrectomy + Nivolumab) (N=357) | Arm B (Nephrectomy Only) (N=377)
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 7 | 9
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1
Asystole (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 3 | 2
Heart failure (Cardiac disorders) | 1 | 0
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1
Myocarditis (Cardiac disorders) | 3 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 1
Death NOS (General disorders) | 1 | 0
Fatigue (General disorders) | 7 | 1
Gait disturbance (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 0
Adrenal insufficiency (Endocrine disorders) | 5 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 6
Colitis (Gastrointestinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 7 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 2
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 2
Obstruction gastric (Gastrointestinal disorders) | 1 | 1
Pancreatic fistula (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 4 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0
Anaphylaxis (Immune system disorders) | 1 | 0
Autoimmune disorder (Immune system disorders) | 2 | 0
Immune system disorders - Other, specify (Immune system disorders) | 4 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Encephalitis infection (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 3
Sepsis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 3 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury to inferior vena cava (Injury, poisoning and procedural complications) | 1 | 0
Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 1
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 10 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 1
Cardiac troponin I increased (Investigations) | 1 | 0
CPK increased (Investigations) | 2 | 0
Creatinine increased (Investigations) | 4 | 1
Lipase increased (Investigations) | 17 | 1
Lymphocyte count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 1 | 0
Serum amylase increased (Investigations) | 9 | 0
Urine output decreased (Investigations) | 1 | 2
Investigations - Other, specify (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 6 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Myelitis (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 2 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 2 | 0
Extraocular muscle paresis (Eye disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 8 | 6
Chronic kidney disease (Renal and urinary disorders) | 1 | 2
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 | 2
Hypertension (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 2 | 3
Peripheral ischemia (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 4 | 6
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Nephrectomy + Nivolumab) (N=357) | Arm B (Nephrectomy Only) (N=377)
Anemia (Blood and lymphatic system disorders) | 30 | 21
Fatigue (General disorders) | 138 | 28
Pain (General disorders) | 16 | 21
Dry skin (Skin and subcutaneous tissue disorders) | 18 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 89 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 89 | 2
Hyperthyroidism (Endocrine disorders) | 18 | 0
Hypothyroidism (Endocrine disorders) | 54 | 0
Abdominal pain (Gastrointestinal disorders) | 29 | 51
Constipation (Gastrointestinal disorders) | 18 | 13
Diarrhea (Gastrointestinal disorders) | 45 | 2
Nausea (Gastrointestinal disorders) | 52 | 24
Alanine aminotransferase increased (Investigations) | 40 | 4
Aspartate aminotransferase increased (Investigations) | 41 | 2
Creatinine increased (Investigations) | 57 | 30
Lipase increased (Investigations) | 25 | 2
Serum amylase increased (Investigations) | 22 | 1
Anorexia (Metabolism and nutrition disorders) | 24 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 19 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT03055013/Prot_SAP_000.pdf